CLINICAL TRIAL: NCT00909467
Title: Early Recognition of Pulmonary Arterial Hypertension in Myelodysplastic and Myeloproliferative Diseases
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 20-097 ex 08/09
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Myeloproliferative Disorder; Myelodysplastic Syndromes; Pulmonary Hypertension
MeSH Terms: conditions — Myeloproliferative Disorders; Myelodysplastic Syndromes; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA will be retained for later examinations at the Department for Genetics, if the patient agrees with it (specific question at the patient information).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- myeloproliferative, -dysplastic disease
  Interventions: Other: echocardiography, right heart catheterisation

INTERVENTIONS:
Other: echocardiography, right heart catheterisation — at each patient an echocardiography will be performed at rest and during exercise. For the evaluation of exercise capacity, cardiopulmonary exercise testing and six-minute walk is performed. Right heart catheterisation is recommended to those with suspected pulmonary hypertension.
  Other Names: EDE, RHC

SUMMARY:
Myelodysplastic and myeloproliferative Disease represent conditions with increased risk for pulmonary hypertension. However, the exact prevalence of pulmonary hypertension in these conditions is not known. The effects of pulmonary hypertension on the clinical picture and the symptoms of patients in these conditions needs also further exploration. This exploratory study is designed to describe the prevalence of pulmonary hypertension in the population with such hematologic diseases, and the stages of pulmonary hypertension as well its effect on exercise capacity at time of diagnosis.

DETAILED DESCRIPTION:
For early recognition of pulmonary hypertension exercise doppler echocardiography will be used in all patients. Patients with elevated pulmonary arterial pressure at rest or during exercise (estimated by echocardiography), or with decreased exercise capacity (as a potential sign of pulmonary hypertension) are advised to undergo right heart catheterisation. Cardiopulmonary exercise testing and six-minute walk distance measurement are performed to measure exercise capacity. The described work-up of patients allows precise and objective hemodynamic and clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* myelodysplastic disease or myeloproliferative diseases

Exclusion Criteria:

* known pulmonary hypertension
* relevant pulmonary disease
* relevant left cardiac or valvular disease
* recent major operations
* recent changes in medications
* relevant anaemia
* inability to exercise

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with known myeloproliferative or myelodysplastic disease as a risk factor for pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
mean pulmonary arterial pressure at rest and during exercise | at baseline and after 1 year

SECONDARY OUTCOMES:
exercise capacity | at baseline and after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz, Pulmonology
Locations (1):
- Medical University of Graz, Pulmonology, Graz, Austria